CLINICAL TRIAL: NCT07049029
Title: Physical Activity Pain Resilience
Acronym: PAPR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: William Black (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor-Investigator, William Black, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00004982; K23AR078337 (NIH)
Record Dates: First submitted 2025-06-13; First posted 2025-07-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain
Keywords: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PREP-Y (Experimental)
  Interventions: Behavioral: PREP-Y

INTERVENTIONS:
Behavioral: PREP-Y — The intervention is a series of behavioral health/psychoeducational modules that the participant will learn from. Participants will use the information discussed and overall impact on physical activity engagement, chronic pain management, and quality of life will be measured

SUMMARY:
The purpose of this research study is to test a new program called Pain REsilience Promotion for Youth (PREP-Y). This program is designed to help adolescents with chronic musculoskeletal pain (pain in muscles, bones, or joints that lasts more than 3 months) become more physically active and better able to manage their pain. The program includes four weekly virtual sessions that teach skills related to resilience, such as how to stay motivated, build confidence, and cope with pain.

Participants will complete surveys and physical activity tests before and after the program. Participants will also wear physical activity monitors to track their activity levels. The goal of this study is to learn whether the program is practical, helpful, and acceptable to participants, and to prepare for a future larger study.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 12 and 17
* History of chronic musculoskeletal pain for more than 3 months assessed by a pediatric rheumatologist or pain physician
* Diagnosis of a primary pain disorder (e.g., juvenile fibromyalgia and other widespread pain conditions, lower back pain, complex regional pain and amplified pain syndrome)
* Speaks English as primary language

Exclusion Criteria:

* Chronic pain secondary to disease (e.g., sickle cell disease or rheumatic disease such as juvenile arthritis, systemic lupus erythematosus)
* Presence of an untreated major psychiatric diagnosis (e.g., major depression, bi-polar disorder, psychoses)
* History or diagnosis of developmental delay.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention | From enrollment to the post-treatment visit, for a total of 6 weeks
  Fidelity checklists detailing content areas of the intervention adequately conveyed during the study visit will be used to measure intervention feasibility.
Acceptability of Intervention | From enrollment to the post-treatment visit, for a total of 6 weeks
  Number of intervention visits completed by participants will be used to determine how acceptable the intervention is to the target population.

SECONDARY OUTCOMES:
Accelerometry Data | From baseline to 3-month follow-up, for a total of 18 weeks
  Activity from the Actigraphs will assist in understanding and identifying changes in participant physical activity.
Functional Disability Inventory | From baseline to 3-month follow-up, for a total of 18 weeks
  The Functional Disability Inventory is a 15-item questionnaire that measures an individual's perception of how their illness limits their ability to complete regular activities. A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: William Black, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided